CLINICAL TRIAL: NCT02194946
Title: Effectiveness of Chinese Medicine on Deferring Dialysis Initiation for Stage 5 Chronic Kidney Disease
Brief Title: Chinese Medicine on Deferring Dialysis Initiation
Acronym: C-MODDI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Liu Xu-sheng, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013BAI02B04
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: End-Stage Renal Disease
Keywords: Chronic Kidney Disease,; End-Stage Renal Disease,; Traditional Chinese Medicine,; dialysis initiation.
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Medicine, Chinese Traditional; Therapeutics; Complementary Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CKD-related management group (Active Comparator): Patients in basic care group are provided with basic western medicine treatment according to Kidney Disease: Improving Global Outcomes(KDIGO) and The National Kidney Foundation Kidney Disease Outcomes Quality Initiative(KDOQI) guidelines but not prescribed any Chinese herbal medicine.
  The basic western medicine treatment mainly includes dietary protein restriction(0.6g/kg·d, for Chinese), Blood pressure control, treating anemia with erythropoietin,treatment of abnormal calcium-phosphate metabolism, and treatment of fluid, electrolyte and acid-base disorders.
  Interventions: Drug: CKD-related management
- CM therapies group (Experimental): Participants will receive CM therapies and CKD-related management concurrently. One or several the following CM patterns will be allowed: a. Chinese herbal formula via oral administration; b. Chinese patent medicine via oral administration; c. Chinese herbal formula via colonic administration; d. Chinese patent medicine via colonic administration.
  Interventions: Drug: CM therapies; Drug: CKD-related management

INTERVENTIONS:
Drug: CM therapies — The choice of CM patterns will be at the treating physician's discretion. The dosing regimen of Chinese herbs and Chinese patent medicine will be as per the 2010 Chinese pharmacopoeia.The oral Chinese herbal formula will be composed of 18 herbs:Radix Astragali, Radix Codonopsis, Rhizoma Atractylodis Macrocephalae, Rhizoma diosscoreae, Poria, Semen Cuscutae, Radix Morindae Officinalis, Herba Epimedii, Herba Cistanches, Fructus Ligustri Lucidi, Rhizoma Polygonati, Fructus Amomi, Herba Agastaches, Rhizoma Coptidis, Radix et Rhizoma Rhei, Semen Coicis, Radix Salviae Miltiorrhizae, and stir-baked Semen Persicae. The Chinese herbal formula via Colonic administration will be composed of 3 herbs: Radix et Rhizoma Rhei, Calcined Concha Osterae, Herba Taraxaci.
  Other Names: Traditional Chinese medicine (TCM) treatment; TCM treatment; Complementary Therapies
  Arms: CM therapies group
Drug: CKD-related management — Western medicine treatment for CKD are practised following KDIGO and KDOQI guidelines, to reach the recommended goals of nutrition, blood pressure, hemoglobulin, electrolytes, fluid control and acid-base balance.
  Other Names: modern medicine; Western medicine

SUMMARY:
Stage 5 chronic kidney disease (CKD), also end stage renal disease(ESRD), usually presents overt clinical symptoms and is a critical stage when patients are encountered with dialysis. The optimal time to initiating dialysis in patients with stage 5 CKD is addressed as the most important dialysis-related question. As indicated by the recently published European Renal Best Practice (ERBP) guideline, early initiation seemed to produce no benefit but greater expenditure and sometimes more harm.Renal replacement therapies (RRT) including dialysis are the most common procedures for patients with end-stage renal disease (ESRD), but conservative management should be an option in patients who still experience the stable period without clinical indications of dialysis.Chinese Medicine (CM) is recognized as an alternative therapy on alleviating uremic symptoms, deferring dialysis initiation, and improving quality of life. Although the effects of CM on kidney disease have been demonstrated in animal experiments, evidence from large clinical trial is insufficient. So we raise the hypothesis that CM therapies including Chinese herbal formula, Chinese patent medicine via oral pattern and/or Colonic administration, will defer the initiation of dialysis in adults with stage 5 CKD.

DETAILED DESCRIPTION:
Chinese Medicine (CM) treatment has been applied to CKD patients commonly in China, especially those independent of dialysis. Based on the personal experience of experts from different areas in China, patients with stage 5 CKD have been treated with different formulations of herbs including Astragalus membranaceus (Huangqi), Codonopsis pilosula (Dangshen), Semen Cuscutae (Tusizi) and Radix et Rhizoma Rhei (Dahuang) etc. . Based on the Traditional Chinese Medicine theory and clinical practise, these herbal medicines help strengthening "spleen-kidney" and dispelling "turbidity" . To determine whether CM therapies including Chinese herbal formula, Chinese patent medicine via oral pattern and/or Colonic administration, will significantly defer dialysis initiation, we conduct the Chinese Medicine on Deferring Dialysis Initiation (C-MODDI) study. It's a multicenter, prospective, controlled trial, also an effectiveness study that are conducted in the "real world" of a variety of busy clinical practices, with heterogeneous interventions that are more representative of the general effectiveness of CM therapies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years;
* with an estimated glomerular filtration rate (eGFR) between 5.5-15 ml/min per 1.73 m2;
* Non-diabetic CKD, which should be identified by biopsy or patients' medical histories.
* East Asian.

Exclusion Criteria:

* Clinical indications of dialysis still occur after conservative kidney management for 1 week, which will be ruled out as hemoglobin < 70g/L; or serum potassium> 6.5mmol/L; or Carbon Dioxide Combining Power (CO2CP) <13mmol/L; or EPI-GFR≤5ml/min/1.73m2 ;
* Pregnant or lactating.
* Critical status, such as alimentary tract hemorrhage or decompensated cirrhosis;
* History of malignancy other than a successfully and completely treated carcinoma;
* Any condition (mental or physical) that would interfere with the patient's ability to comply with the study protocol;
* Concurrent or current treatment with glucocorticoid or immunosuppressant agents in last 3 months;
* Participation in any other clinical trial;
* Known or suspected allergy to certain agents involved;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 875 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to initiation of dialysis from enrollment. | From enrollment to dialysis initiation or death.The duration of follow up will be for a maximum of 4 years.
  Averaged time from enrollment to dialysis initiation or death from any cause, whichever comes first.
  Patients commence dialysis based on the following criteria:
  1. Clinical indications of dialysis include medically refractory serum potassium> 6.5mmol/L, total carbon dioxide (TCO2) <13mmol/L, eGFR≤5ml/min/1.73m2 (calculated by EPI formula), or the patient is symptomatic (see criteria #2). If these indications remain occur after receiving conservative CKD-related management for 1 week, or if relapse twice within one month, the patient definitely reaches the endpoint.
  2. Uremic symptoms include nausea, vomit, malnutrition, pericarditis or pleurisy, volume overload, encephalopathy, bleeding tendency, refractory hypertension, or other symptoms that are likely to be ameliorated by dialysis.

SECONDARY OUTCOMES:
all-cause mortality | From enrollment to dialysis initiation or death.The duration of follow up will be for a maximum of 4 years.
  percentage of subjects who die from any cause during follow-up.
Cardio-cerebro vascular events | From enrollment to dialysis initiation or death.The duration of follow up will be for a maximum of 4 years.
  Cardio-cerebro vascular events, i.e. cerebral hemorrhage, cerebral infarction, myocardial infarction, acute coronary syndrome, severe arrhythmia, acute heart failure, acute exacerbation of congestive heart failure.
Hospitalization or death caused by severe infection. | From enrollment to dialysis initiation or death.The duration of follow up will be for a maximum of 4 years.
  percentage of subjects who suffer from severe infection events before dialysis initiation.The severe infection will lead to hospitalization or death.
  Infection events refer to death or hospitalization due to infection.
incidence of severe adverse event/reaction | From enrollment to dialysis initiation or death.The duration of follow up will be for a maximum of 4 years.
  number of cases of any recorded severe adverse event/reaction per year. Any adverse events/reactions complained of by patients or observed by researchers should be recorded, as well as any newly accompanied disease or aggravation of original symptoms.
Slope of reciprocal serum creatinine | From date of enrollment until the date of first dialysis or date of death from any cause,or the end of study, whichever come first.The duration of follow up will be for a maximum of 4 years.
  Reciprocal serum creatinine (1/SCr) slope,the serum creatinine was assessed every 2 months.
Nutrition and microinflammation status | From date of enrollment until the date of death from any cause,or the end of study, whichever come first, performed every 6 months.The duration of follow up will be for a maximum of 4 years.
  Malnutrition Inflammation Score is used to assess nutrition and microinflammation status.

OTHER OUTCOMES:
Liver function | From date of enrollment until the date of death from any cause,or the end of study, whichever come first, performed every 6 months.The duration of follow up will be for a maximum of 4 years.
  aspartate aminotransferase (AST),alanine aminotransferase (ALT)
Complete blood count | From date of enrollment until the date of death from any cause,or the end of study, whichever come first, performed every 6 months.The duration of follow up will be for a maximum of 4 years.
  Complete blood count
Routine stool test + occult blood | From date of enrollment until the date of death from any cause,or the end of study, whichever come first, performed every 6 months.The duration of follow up will be for a maximum of 4 years.
  Routine stool test + occult blood
Electrocardiogram | From date of enrollment until the date of death from any cause,or the end of study, whichever come first, performed every 6 months.The duration of follow up will be for a maximum of 4 years.
  Electrocardiogram
Adverse event/reaction | From date of enrollment until the date of death from any cause,or the end of study, whichever come first, performed every 6 months.The duration of follow up will be for a maximum of 4 years.
  number of cases of any recorded adverse event/reaction per year.

CONTACTS AND LOCATIONS:
Overall Officials: Xusheng Liu, MD, Study Director — Guangdong Provincial Hospital of Traditional Chinese Medicine; Ping Li, PhD, Principal Investigator — China-Japan Friendship Hospital
Locations (29):
- China (29):
  - Anhui Provincial Hospital of Chinese Medicine, Hefei, Anhui
  - China PLA General Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Dongzhimen Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - First Hospital of Peking University, Beijing, Beijing Municipality
  - Guang'anmen Hospital China Academy of traditional Chinese Medicine, Beijing, Beijing Municipality
  - Xiyuan Hospital, Academy of traditional Chinese Medicine, Beijing, Beijing Municipality
  - Third Military Medical University Xinqiao Hospital, Chongqing, Chongqing Municipality
  - General hospital of Guangzhou Military command of PLA, Guangzhou, Guangdong
  - Guangzhou No.1 People's Hospital, Guangzhou, Guangdong
  - Huadu District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - TCM Integrated Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Liuzhou Hospital of traditional Chinese Medicine, Liuchow, Guangxi
  - First Affiliated Hospital of Guangxi University Of Chinese Medicine, Nanning, Guangxi
  - First Affiliated Hospital of Guiyang College of Traditional Chinese Medicine, Guiyang, Guizhou
  - First Affiliated Hospital of Heilongjiang University Of Chinese Medicine, Harbin, Heilongjiang
  - Heilongjiang Academy of Traditional Chinese Medicine, Harbin, Heilongjiang
  - Hubei Provincial Hospital of Chinese Medicine, Wuhan, Hubei
  - Jiangsu Provincial Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Shaanxi Provincial Hospital of Chinese Medicine, Xi'an, Shaanxi
  - Xijing Hospital of The Fourth Military Medical University, Xi'an, Shaanxi
  - Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - The Sixth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - First hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - First Affiliated Hospital of Tianjin University Of Chinese Medicine, Tianjin, Tianjin Municipality
  - Hangzhou Hospital of Chinese Medicine, Hangzhou, Zhejiang
  - Tong De Hospital, Zhejiang Province, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wang YJ, He LQ, Sun W, Lu Y, Wang XQ, Zhang PQ, Wei LB, Cao SL, Yang NZ, Ma HZ, Gao J, Li P, Tao XJ, Yuan FH, Li J, Yao C, Liu X. Optimized project of traditional Chinese medicine in treating chronic kidney disease stage 3: a multicenter double-blinded randomized controlled trial. J Ethnopharmacol. 2012 Feb 15;139(3):757-64. doi: 10.1016/j.jep.2011.12.009. Epub 2011 Dec 13. PMID 22178174
- [Background] Zou C, Lu ZY, Wu YC, Yang LH, Su GB, Jie XN, Liu XS. Colon may provide new therapeutic targets for treatment of chronic kidney disease with Chinese medicine. Chin J Integr Med. 2013 Feb;19(2):86-91. doi: 10.1007/s11655-013-1351-8. Epub 2013 Jan 31. PMID 23371456
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD Work Group. KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. Kidney inter., Suppl.2013;3: 1-150.
- [Background] Rosansky S, Glassock RJ, Clark WF. Early start of dialysis: a critical review. Clin J Am Soc Nephrol. 2011 May;6(5):1222-8. doi: 10.2215/CJN.09301010. PMID 21555505
- [Background] Rosansky SJ, Clark WF, Eggers P, Glassock RJ. Initiation of dialysis at higher GFRs: is the apparent rising tide of early dialysis harmful or helpful? Kidney Int. 2009 Aug;76(3):257-61. doi: 10.1038/ki.2009.161. Epub 2009 May 20. PMID 19455195
- [Background] Wright S, Klausner D, Baird B, Williams ME, Steinman T, Tang H, Ragasa R, Goldfarb-Rumyantzev AS. Timing of dialysis initiation and survival in ESRD. Clin J Am Soc Nephrol. 2010 Oct;5(10):1828-35. doi: 10.2215/CJN.06230909. Epub 2010 Jul 15. PMID 20634325
- [Background] Rosansky SJ, Eggers P, Jackson K, Glassock R, Clark WF. Early start of hemodialysis may be harmful. Arch Intern Med. 2011 Mar 14;171(5):396-403. doi: 10.1001/archinternmed.2010.415. Epub 2010 Nov 8. PMID 21059968
- [Background] Hwang SJ, Yang WC, Lin MY, Mau LW, Chen HC; Taiwan Society of Nephrology. Impact of the clinical conditions at dialysis initiation on mortality in incident haemodialysis patients: a national cohort study in Taiwan. Nephrol Dial Transplant. 2010 Aug;25(8):2616-24. doi: 10.1093/ndt/gfq308. Epub 2010 Jun 2. PMID 20519231
- [Background] Cooper BA, Branley P, Bulfone L, Collins JF, Craig JC, Fraenkel MB, Harris A, Johnson DW, Kesselhut J, Li JJ, Luxton G, Pilmore A, Tiller DJ, Harris DC, Pollock CA; IDEAL Study. A randomized, controlled trial of early versus late initiation of dialysis. N Engl J Med. 2010 Aug 12;363(7):609-19. doi: 10.1056/NEJMoa1000552. Epub 2010 Jun 27. PMID 20581422
- [Background] Nesrallah GE, Mustafa RA, Clark WF, Bass A, Barnieh L, Hemmelgarn BR, Klarenbach S, Quinn RR, Hiremath S, Ravani P, Sood MM, Moist LM; Canadian Society of Nephrology. Canadian Society of Nephrology 2014 clinical practice guideline for timing the initiation of chronic dialysis. CMAJ. 2014 Feb 4;186(2):112-7. doi: 10.1503/cmaj.130363. No abstract available. PMID 24492525
- [Background] Tattersall J, Dekker F, Heimburger O, Jager KJ, Lameire N, Lindley E, Van Biesen W, Vanholder R, Zoccali C; ERBP Advisory Board. When to start dialysis: updated guidance following publication of the Initiating Dialysis Early and Late (IDEAL) study. Nephrol Dial Transplant. 2011 Jul;26(7):2082-6. doi: 10.1093/ndt/gfr168. Epub 2011 May 5. No abstract available. PMID 21551086
- [Background] Li Z, Zhu L, Zhang H, Yang J, Zhao J, Du D, Meng J, Yang F, Zhao Y, Sun J. Protective effect of a polysaccharide from stem of Codonopsis pilosula against renal ischemia/reperfusion injury in rats. Carbohydr Polym. 2012 Nov 6;90(4):1739-43. doi: 10.1016/j.carbpol.2012.07.062. Epub 2012 Jul 31. PMID 22944441
- [Background] Song J, Meng L, Li S, Qu L, Li X. A combination of Chinese herbs, Astragalus membranaceus var. mongholicus and Angelica sinensis, improved renal microvascular insufficiency in 5/6 nephrectomized rats. Vascul Pharmacol. 2009 May-Jun;50(5-6):185-93. doi: 10.1016/j.vph.2009.01.005. PMID 19563735
- [Background] Tong Y, Han B, Guo H, Liu Y. Protection of Chinese herbs against adenine-induced chronic renal failure in rats. Afr J Tradit Complement Altern Med. 2010;7(4):331-8. doi: 10.4314/ajtcam.v7i4.56701. Epub 2010 Jul 3. PMID 21731165
- [Background] Chinese Pharmacopoeia Commission. Pharmacopoeia of the People's Republic of China. Beijing: People's Medicial Publishing House; 2010
- [Background] Emmanuel AV, Krogh K, Bazzocchi G, Leroi AM, Bremers A, Leder D, van Kuppevelt D, Mosiello G, Vogel M, Perrouin-Verbe B, Coggrave M, Christensen P; Members of working group on Trans Anal Irrigation from UK, Denmark, Italy, Germany, France and Netherlands. Consensus review of best practice of transanal irrigation in adults. Spinal Cord. 2013 Oct;51(10):732-8. doi: 10.1038/sc.2013.86. Epub 2013 Aug 20. PMID 23958927